CLINICAL TRIAL: NCT02011217
Title: The Effects of Rye Crisp Bread on Subjective Appetite and Metabolic Function After Short-term Consumption
Brief Title: The Effects of Rye Crisp Bread on Appetite and Metabolic Function
Acronym: S2RBAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swedish University of Agricultural Sciences (Other)
Collaborators: Uppsala University (Other)
Responsible Party: Principal Investigator, Isabella Lee, PhD student, Swedish University of Agricultural Sciences
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: SLU-IL-S2
Record Dates: First submitted 2013-11-06; First posted 2013-12-13 (Estimated); Last update posted 2013-12-13 (Estimated); Status verified 2013-12

CONDITIONS: Appetite Regulation
Keywords: Rye; Dietary Fibre; Bread; Crisp bread; Appetite; Satiety; Hunger; Desire to eat; Metabolism; Glucose; Insulin; Gut hormones; Gastric emptying rate
MeSH Terms: conditions — Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rye crisp bread A (Experimental)
  Interventions: Other: Rye crisp bread B; Other: Wheat crisp bread C
- Rye crisp bread B (Experimental)
  Interventions: Other: Rye crisp bread A; Other: Wheat crisp bread C
- Wheat crisp bread C (Experimental)
  Interventions: Other: Rye crisp bread A; Other: Rye crisp bread B

INTERVENTIONS:
Other: Rye crisp bread A — In a randomized cross-over design each subject receive one of three iso-caloric breakfasts on three different occasions, separated by 1 week wash-out period.
  Arms: Rye crisp bread B; Wheat crisp bread C
Other: Rye crisp bread B — In a randomized cross-over design each subject receive one of three iso-caloric breakfasts on three different occasions, separated by 1 week wash-out period.
  Arms: Rye crisp bread A; Wheat crisp bread C
Other: Wheat crisp bread C — In a randomized cross-over design each subject receive one of three iso-caloric breakfasts on three different occasions, separated by 1 week wash-out period.
  Arms: Rye crisp bread A; Rye crisp bread B

SUMMARY:
The aim of this study is to contribute to a better understanding of how dietary fibre in rye affects appetite and metabolic processes. We will evaluate how the intake of rye crisp breads affects appetite, insulin secretion and glucose levels in the blood in healthy humans. We will also investigate microstructural properties of the crisp breads with microscopy, as well as to characterize the food products with respect to the content of dietary fibre and certain bioactive compounds. The aim is also to try to elucidate how observed effects on appetite are related to changes in insulin and glucose levels, appetite related hormonal signals and microstructural properties to verify findings from previous studies.

DETAILED DESCRIPTION:
The short-term effects (up to 4 hours after intake) of rye crisp breads on subjective appetite and metabolism will be evaluated using a randomized cross-over study design. Each participant will consume three different breakfasts consisting of two different rye crisp breads and one wheat crisp bread on three different occasions separated by a 1 week wash-out period. Participants will rate subjective appetite (satiety, hunger and desire to eat) by using a visual analogue scale (VAS) every 30 min during a 4-hour period, starting 30 min before breakfast. Blood samples will be collected before breakfast and at regular intervals throughout the day for analysis of glucose, insulin and hormone levels. Gastric emptying rate will also be evaluated using paracetamol as an indicator. Glucose and hormonal responses will be related to subjective appetite and to differences in composition of the breakfasts.

ELIGIBILITY:
Inclusion Criteria:

* Habitual breakfast eaters

Exclusion Criteria:

* Pregnancy, lactation or wishing to become pregnant during the study period
* Dieting
* Weightloss
* Eating disorder
* Hyperglycemic
* Hyperinsulinemic
* Thyroid disease
* Metabolic issues
* Diabetes
* Physical or psychological problems with eating
* Food intolerance/allergies to foods included in the study
* Intolerance/allergy to paracetamol
* Heavy smokers
* Recent or concurrent participation in a dietary intervention research study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-08; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Subjective Appetite Profiles during 4 hours | -30, 0, 30, 60, 90, 120, 150, 180, 210, 240 minutes
  Subjective feelings of appetite (satiety, hunger and desire to eat) assessed by visual analogue scale (VAS).

SECONDARY OUTCOMES:
Gastric Emptying Rate during 4 hours | -15, 15, 35, 65, 95, 125, 185, 230 minutes
  Paracetamol (1 g) taken with breakfast. The appearance of paracetamol in the blood is directly related to the rate of gastric emptying.
Hormonal Responses during 4 hours | -15, 15, 35, 65, 95, 125, 185, 230 minutes
  Glucagon, glucagon-like peptide-1 (GLP-1), glucose-dependent insulino-tropic polypeptide (GIP), peptide YY (PYY), cholecystokinin (CCK), leptin and ghrelin are measured in plasma samples.
Glucose and Insulin Responses during 4 hours | -15, 15, 35, 65, 95, 125, 185, 230 minutes
  Glucose and insulin are measured in plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Rikard K Landberg, Ass. Prof., Principal Investigator — Swedish University of Agricultural Sciences
Locations (1):
- Paediatric Research Facility; The Children's Hospital at Uppsala University Hospital, Uppsala, Uppsala County, Sweden

REFERENCES:
- [Derived] Johansson DP, Lee I, Riserus U, Langton M, Landberg R. Effects of unfermented and fermented whole grain rye crisp breads served as part of a standardized breakfast, on appetite and postprandial glucose and insulin responses: a randomized cross-over trial. PLoS One. 2015 Mar 31;10(3):e0122241. doi: 10.1371/journal.pone.0122241. eCollection 2015. PMID 25826373